CLINICAL TRIAL: NCT04594421
Title: Study on the Increasing Proportion and Change Trend of Eosinophil in Peritoneal Fluid During Peritoneal Dialysis-Related Peritonitis
Brief Title: Change Trend of Effluent Eosinophil During Peritoneal Dialysis-Related Peritonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Professor in Renal Divison,Department of Medicine, Peking University First Hospital
Other Study IDs: Eosinophil increase
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Peritonitis
Keywords: Peritonitis; eosinophil; peritoneal dialysis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multi-center prospective cohort study will be conducted to explore the change trend of eosinophil in peritoneal dialysis effluent during peritoneal dialysis-associated peritonitis, and to explore the relationship between eosinophil increase, peritonitis severity and antibiotic use. This study will provide evidence for routine eosinophil testing

DETAILED DESCRIPTION:
A multi-center prospective cohort study will be conducted to explore the change trend of eosinophil in peritoneal dialysis effluent during peritoneal dialysis-associated peritonitis, and to explore the relationship between eosinophil increase, peritonitis severity and antibiotic use. In this study, 100 patients with peritoneal dialysis-associated peritonitis who meet the inclusion criteria will be selected. Demographic data, laboratory variables, peritoneal fluid cytology and bacterial culture will be collected within 24 hours of peritonitis (day 1). Peritoneal fluid cytology includes leukocyte classification and eosinophilic leukocyte count will be examined at day 3, 5, 7, 10, 14, 21, 30, 60 and 90 after peritonitis. All patients will be followed up for 90 days, and their peritonitis outcome will be recorded. The primary endpoint is the prevalence of eosinophil increase in peritoneal effluent, which is defined as >100 eosinophils/mm^3, or >10% eosinophils of the total non-erythrocyte count. Secondary end points are peritonitis outcome at month 1 and 3 including transfer to hemodialysis , death.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as peritoneal dialysis-related peritonitis;
* Age> 14 years
* Maintenance peritoneal dialysis due to end-stage renal failure ≥3 months
* Use of lactate glucose dialysate

Exclusion Criteria:

* Those who cannot be followed up regularly
* Reluctant to join this researcher

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients on peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of elevated eosinophils in peritoneal dialysis effluent | Feb 18,2021 to December 31,2023
  eosinophil number >100 /mm3, or the proportion of polynuclear leukocytes >10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Division and Institute of Nehprology,Peking University First Hospital, Beijing, Beijing Municipality, China